CLINICAL TRIAL: NCT00933660
Title: Do we Need an Instructor, or a Manikin to Learn BLS/AED, or is Web Based Training as Good as Instructor Based Training?
Brief Title: Retention and Retrieval for Three Different Training Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Doczero (Other)
Collaborators: Ambulance Oost (Unknown)
Responsible Party: Wiebe de Vries, Doczero
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 081203_Ed-web
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Improvement of BLS/AED Training Methods
Keywords: Education; Retention; Retrieval

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control-1 (Active Comparator): ERC-training by instructor
  Interventions: Other: ERC-training by instructor
- Control-2 (No Intervention): No intervention
- Experimental-1 (Experimental): Web-based training only
  Interventions: Other: Web-based training only
- Experimental-2 (Experimental): Web-based training with a personal training manikin
  Interventions: Other: Web-based training with a personal training manikin

INTERVENTIONS:
Other: ERC-training by instructor — Standard way of training with an instructor
  Arms: Control-1
Other: Web-based training only — Experimental way of training with a web based training application
  Arms: Experimental-1
Other: Web-based training with a personal training manikin — Experimental way of training with a web based training application and a simple personal training manikin
  Arms: Experimental-2

SUMMARY:
The hypotheses that will be studied are:

H0: Providers trained by a web based application for skill competency in basic life support (BLS) and automated external defibrillation (AED) are as competent as those who were trained by certified instructors using the European Resuscitation Council (ERC) curriculum

H00-1: Providers who trained themselves with the used of web based training are more competent when they had a personal manikin for home exercise compared to providers who trained themselves with only a web based training

H0-2: Providers who did not receive any training will score lower than those who did.

Research questions for this study are:

1. What are the results in skill competency for non trained people?
2. What are the results in skill competency for trained people immediately after training?
3. What is the retention of skills for trained and non trained people after six months?

ELIGIBILITY:
Inclusion Criteria:

* willing to follow a BLS/AED course

Exclusion Criteria:

* CPR training within the last five years
* professional health care provider

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-03 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Kruskal-Wallis | 10-2007 - 03-2009

CONTACTS AND LOCATIONS:
Overall Officials: Wiebe de Vries, MSc, Principal Investigator — Doczero; Koenraad Monsieurs, Professor, Study Chair — University Hospital, Ghent; Joost Bierens, Professor, Study Director — VU Medical Centre; Rudolph Koster, PhD, Study Chair — Academical Medical Centre Amsterdam